CLINICAL TRIAL: NCT05168488
Title: Repeatability of Blood Glucose Responses to Fasted and Fed Resistance Exercise in Individuals With Type 1 Diabetes
Brief Title: Repeatability of Blood Glucose Responses to Resistance Exercise in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00082031
Record Dates: First submitted 2021-11-22; First posted 2021-12-23 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): There is only one study arm consisting of all participants.
  Interventions: Behavioral: Fasted morning resistance exercise; Behavioral: Afternoon resistance exercise

INTERVENTIONS:
Behavioral: Fasted morning resistance exercise — On three separate occasions, participants will perform a standardized resistance exercise protocol in the morning while fasting.
Behavioral: Afternoon resistance exercise — On three separate occasions participants will perform a standardized resistance exercise protocol in the afternoon after eating their regular lunch

SUMMARY:
This study proposes to examine the impact of time of day (morning versus afternoon) on the variability of blood glucose responses to high resistance exercise in a single group of patients with type 1 diabetes. Participants will be asked to wear a continuous glucose monitor during the 3 weeks of testing. During the six exercise sessions (three in the morning while fasted and three in the afternoon), participants will complete the same resistance exercise protocol.

DETAILED DESCRIPTION:
Pre-test measures: Interested participants will be invited to the Physical Activity and Diabetes Laboratory on the main campus of the University of Alberta. They will be asked questions related to their physical activity levels and medication, and blood pressure will be measured to assess their eligibility. Where participants are eligible, anthropometric characteristics will be measured using standard protocols, as will blood pressure. A blood sample will be drawn for assessment of HbA1c. Participants will be introduced to the weight lifting equipment and the proper lifting techniques associated with each exercise prior to performing a standardized test to determine the maximum weight they can safely lift eight times while maintaining proper form (8 repetition maximum - 8RM).

Testing sessions: Participants will be asked to arrive at the lab either between 7 and 8 am in a fasting state, or between 4 pm and 5 pm. The three morning and three afternoon testing sessions will have identical exercise protocols. Participants will be asked to perform three sets of eight repetitions of seven different exercises (bench press leg press, shoulder press, leg curl, lat pulldown, abdominal crunches, seated row) at their pre-determined 8RM. Participants will be asked to match their food and insulin intake as closely as possible on testing days to avoid having these as confounders.

A continuous glucose monitor (CGM) sensor will be subcutaneously inserted by one of the investigators (trained by a group from the CGM manufacturer) into the anterior abdominal area of the participant in the morning of the day prior to the first testing session. CGM will store glucose data every 5 minutes for up to 7 days. During this time, participants will be asked to wear an accelerometer to allow for the objective assessment of background physical activity and sleep quality. Along with this device, they will fill out an activity and sleep log to improve the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes diagnosed for at least 1 year
* aged 18 to 55 years

Exclusion Criteria:

* HbA1c > 9.9%
* frequent and unpredictable hypoglycemia
* change in insulin management strategy within two months of study
* using closed-loop insulin delivery
* injuries that would contraindicate resistance exercise
* blood pressure > 140/95
* severe peripheral neuropathy
* a history of cardiovascular disease
* severe proliferative retinopathy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
Capillary glucose (change during exercise) | 0 minutes (exercise start), 15 minutes, 30 minutes, 45 minutes, 60 minutes, 75 minutes, 90 minutes
  Using test strips and a hand-held glucometer to test blood from a finger poke

SECONDARY OUTCOMES:
Mean CGM glucose | 6 hours, 12 hours, overnight (midnight to 6am) and 24 hours post-exercise
  mean CGM glucose
CGM coefficient of variation (CV) | 6 hours, 12 hours, overnight (midnight to 6am) and 24 hours post-exercise
  coefficient of variation of continuous glucose monitoring data
CGM standard deviation (SD) | 6 hours, 12 hours, overnight (midnight to 6am) and 24 hours post-exercise
  Standard deviation of CGM glucose
frequency of hypoglycemia | 6 hours, 12 hours, overnight (midnight to 6am) and 24 hours post-exercise
  number of hypoglycemic events measured by CGM
frequency of hyperglycemia | 6 hours, 12 hours, overnight (midnight to 6am) and 24 hours post-exercise
  number of hyperglycemic events measured by CGM
percent time in range | 6 hours, 12 hours, overnight (midnight to 6am) and 24 hours post-exercise
  percent of time spent between 4.0 and 9.9 mmol/L
percent time in hyperglycemia | 6 hours, 12 hours, overnight (midnight to 6am) and 24 hours post-exercise
  percent of time spent over 10.0 mmol/L
percent time in hypoglycemia | 6 hours, 12 hours, overnight (midnight to 6am) and 24 hours post-exercise
  percent of time spent below 3.9 mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Diabetes Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No